CLINICAL TRIAL: NCT01127451
Title: A Phase II Open-Label, Multicenter Study of Denileukin Diftitox in Patients With Stage IIIC and Stage IV Melanoma
Brief Title: Study of Denileukin Diftitox in Participants With Stage IIIC and Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: PharmaBio Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7272-701
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Stage IIIC Melanoma; Stage IV Melanoma
Keywords: Neoplasms
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Denileukin Diftitox on Days 1 to 4 (Experimental): Participants received Denileukin Diftitox 12 mcg/kg/day (microgram per kilogram) on Days 1 through 4 of each 21-day treatment cycle, for a total of 4 cycles (12 weeks).
  Interventions: Drug: Denileukin diftitox
- Denileukin Diftitox on Days 1, 8, and 15 (Experimental): Participants received Denileukin Diftitox 12 mcg/kg/day on Days 1, 8, and 15 of each 21-day treatment cycle, for a total of 4 cycles (12 weeks).
  ARM 2 was closed. Participants experiencing clinical benefit (irSD, irPR, or irCR per irRC) after 4 cycles of treatment, may continue their denileukin diftitox treatment for up to 8 cycles.
  Interventions: Drug: Denileukin diftitox

INTERVENTIONS:
Drug: Denileukin diftitox — Denileukin diftitox intravenous infusion over 30-60 minutes.

SUMMARY:
The purpose of this study is to determine whether participants with Stage IIIC and Stage IV Melanoma experience benefit when treated with Denileukin diftitox in two different dosing schedules.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose/schedule and clinical efficacy study in participants with Stage IIIC and Stage IV melanoma.

Dose-Schedules: This is a schedule, dose, and pharmacodynamic study of Denileukin diftitox in participants with Stage IIIC and Stage IV melanoma. Two arms of 40 participants each were originally planned (see below) for a total of 80 participants. Participants were randomly assigned to 1 of 2 arms: 1. 12 mcg/kg/day on Days 1 through 4 of each 21-day treatment cycle, for a total of 4 cycles (12 weeks); 2. 12 mcg/kg/day on Days 1, 8, and 15 of each 21-day treatment cycle, for a total of 4 cycles (12 weeks). Participants will be evaluated for (clinical response, safety and tolerability, and pharmacodynamic measures of ONTAK activity. An optional substudy will be conducted that will involve collection of serial tumor biopsies at study entry and Day 84 in order to assess tissue pharmacodynamic markers of ONTAK activity (Treg depletion in tumor, appearance of melanoma antigen-specific CD8+lymphocytes, and other markers of mucosal immunity and inflammatory response).

Following an amendment, participants will be enrolled in Arm 1 only (expanded to a total of 55 participants) and Arm 2 was closed. According to the original design, if two responses or less were observed among 22 participants on either arm, that arm would be discontinued.

Participants experiencing clinical benefit (immune-related stable disease [irSD], immune-related partial response [irPR], or immune-related complete response [irCR] per irRC) after 4 cycles of treatment, may continue their denileukin diftitox treatment for up to 8 cycles.

ELIGIBILITY:
Inclusion Criteria Participants may be entered in the study only if they meet all of the following criteria.

1. Male or female participants greater than or equal to18 years of age;
2. Participants with histologically confirmed melanoma (Stage IIIC or Stage IV, American Joint Commission on Cancer);
3. Naive to prior systemic chemotherapy, targeted therapy (eg, BRAF), or immunotherapy (eg, interleukin-2 [IL-2] or interferon) for the treatment of melanoma, including any cytotoxic agents or IL-2 used for adjuvant therapy (adjuvant interferon is allowed). Prior granulocyte macrophage colony-stimulating factor (GM-CSF) is allowed;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2;
5. Life expectancy greater than or equal to 3 months;
6. At least 1 site of radiographically measurable disease by immune-related response criteria (irRC);
7. Serum albumin greater than or equal to 3 g/dL;
8. Adequate hematologic, renal, and liver function as defined by laboratory values performed within 21 days prior to initiation of dosing:

   * Absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L;
   * Platelet count greater than or equal to 100 x 10^9/L;
   * Hemoglobin greater than or equal to 9 g/dL;
   * Serum creatinine less than or equal 1.5 x upper limit of normal (ULN) or creatinine clearance greater than or equal to 50 mL/min;
   * Total serum bilirubin less than or equal to 1.5 x ULN;
   * Serum aspartate transaminase (AST/SGOT) or serum alanine transaminase (ALT/SGPT) less than or equal to 2.5 x ULN, and less than or equal to 5 x ULN if liver metastases are present.
9. Fertile males should use an effective method of contraception during treatment and for at least 3 months after completion of treatment, as directed by their physician;
10. Pre-menopausal females and females less than 2 years after the onset of menopause should have a negative pregnancy test at Screening. Pre-menopausal females must agree to use an acceptable method of birth control from the time of the negative pregnancy test up to 90 days after the last dose of study drug. Females of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for greater than or equal to 1 year; Before study entry, written informed consent must be obtained from the participants prior to performing any study-related procedures.

Exclusion Criteria

Participants will not be entered in the study for any of the following:

1. Known central nervous system (CNS) lesions, except for asymptomatic non-progressing, treated brain metastases.

   Treated brain metastases are defined as having no evidence of progression or hemorrhage for 2 months, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computerized tomography [CT]) during the Screening period (using the pretreatment brain image as Baseline). Treatment for brain metastases must have been completed at least 2 months prior to Day 1 of the first treatment cycle and may include whole brain radiotherapy, radiosurgery (Gamma Knife, LINAC, or equivalent), or a combination as deemed appropriate by the treating physician. Dexamethasone must be discontinued at least 4 weeks prior to Day 1. Participants with CNS metastases treated by neurosurgical resection or brain biopsy performed within 2 months prior to Day 1 will be excluded;
2. Carcinomatous meningitis;
3. Prior treatment with denileukin diftitox;
4. Known hypersensitivity to denileukin diftitox or any of its components: diphtheria toxin, IL-2, or excipients;
5. Prior surgery for melanoma less than 4 weeks before enrollment;
6. Other malignancy within 3 years of randomization, with the exception of adequately treated carcinoma in situ of the cervix or non-melanoma skin cancer, with no subsequent evidence of recurrence and/or malignancies diagnosed at a stage where definitive therapy results in near certain cures. The Medical Monitor must be consulted in such cases;
7. Currently receiving any other anticancer treatment for melanoma (including palliative radiotherapy);
8. Received treatment in another clinical study within the 4 weeks prior to commencing study treatment or participants who have not recovered from side effects of an investigational drug to Common Terminology Criteria for Adverse Events (CTCAE) Grade less than or equal to 1, except for alopecia;
9. Received radiotherapy for non-CNS disease within the 2 weeks prior to commencing study treatment or have not recovered from side effects of all radiation-related toxicities to Grade less than or equal to 1, except for alopecia;
10. Significant cardiovascular impairment (history of congestive heart failure New York Heart Association [NYHA] Grade greater than 2 [see Appendix 5], unstable angina, or myocardial infarction within the past 6 months, or serious cardiac arrhythmia);
11. Use of chronic systemic steroids (>5 days) within 2 weeks of Day 1 of the first treatment cycle (replacement therapy for adrenal insufficiency is allowed);
12. Participants with an allograft requiring immunosuppression;
13. Known positive human immunodeficiency virus (HIV), known hepatitis B surface antigen, or hepatitis C positive;
14. Pregnant, breast-feeding, or refusing double barrier contraception, oral contraceptives, or avoidance of pregnancy measures; Have any other uncontrolled infection or medical condition that could interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-06-22 (Actual); Primary Completion 2015-04-07 (Actual); Study Completion 2015-04-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Encinitas, California
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Chicago, Illinois
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Detroit, Michigan
  - Lincoln, Nebraska
  - Portland, Oregon
  - Amarillo, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 investigative sites in the United States from 22 June 2010 to 07 April 2015.
Pre-assignment Details: A total of 75 participants were randomized and treated.
Groups:
- Denileukin Diftitox on Days 1 to 4: Participants received Denileukin Diftitox 12 microgram per kilogram per day (mcg/kg/day) on Days 1 to 4 of 21-day treatment cycle for a total of 4 cycles (12 weeks) or until unacceptable toxicity or rapid and life-threatening progressive disease.
- Denileukin Diftitox on Days 1, 8, and 15: Participants received Denileukin Diftitox 12 mcg/kg/day on Days 1, 8 and 15 of 21-day treatment cycle for a total of 4 cycles (12 weeks) or until unacceptable toxicity or rapid and life-threatening progressive disease.
Period: Overall Study
Arm/Group | Denileukin Diftitox on Days 1 to 4 | Denileukin Diftitox on Days 1, 8, and 15
Started | 43 | 32
Safety Analysis Set | 43 | 32
Modified Intent-to-Treat (MITT) | 42 | 32
Completed | 0 | 0
Not Completed | 43 | 32
Not completed — Other | 2 | 1
Not completed — Completed 1 Year Follow-up after last dose of study drug | 14 | 12
Not completed — Death | 22 | 17
Not completed — Lost to Follow-up | 3 | 0
Not completed — Administrative Reason by Sponsor | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants enrolled and randomized to treatment and who had any safety assessment following the first dose of study drug.
Groups:
- Denileukin Diftitox on Days 1 to 4: Participants received Denileukin Diftitox 12 mcg/kg/day on Days 1 to 4 of 21-day treatment cycle for a total of 4 cycles (12 weeks) or until unacceptable toxicity or rapid and life-threatening progressive disease.
- Total: Total of all reporting groups
Arm/Group | Denileukin Diftitox on Days 1 to 4 | Denileukin Diftitox on Days 1, 8, and 15 | Total
Number analyzed (Participants) | 43 | 32 | 75
Age, Continuous [Median (Full Range); unit: years] | 66 [38 to 93] | 68 [28 to 94] | 66 [28 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 32 | 20 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 31 | 71
  Asian | 2 | 0 | 2
  Black or African American | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Immune-related Overall Response Rate (irORR)
Description: irORR was defined as the percentage of participants with best confirmed response (immune-related complete response [irCR] or immune-related partial response [irPR]). irORR was assessed by immune-related response criteria (irRC). Per irRC criteria, irCR was defined as complete disappearance of all tumor lesions, whether measurable or not, and no new lesions. irPR was defined as decrease in tumor burden by 50 percent (%) or greater (confirmed in 2 observations at least 4 weeks apart).
Time Frame: From the start of treatment up to 1 year 6 months
Population: MITT included all participants enrolled and randomized to treatment and had an efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Denileukin Diftitox on Days 1 to 4 | Denileukin Diftitox on Days 1, 8, and 15
Number analyzed (Participants) | 42 | 32
percentage of participants | 9.5 [3.3 to 20.4] | 3.1 [0.1 to 13.9]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The PFS was defined as time from start of study treatment until immune-related progressive disease (irPD) or death. If the participant did not progress, the participant was censored at the date of last tumor assessment, known alive, or until starting a next line of therapy, whichever occurred first. PFS was assessed by irRC. irPD was defined as at least 25% increase in tumor burden relative to nadir (at any single time point) in 2 consecutive observations at least 4 weeks apart. The PFS was estimated using the Kaplan-Meier method. The median time (weeks) and the corresponding 90% confidence interval were estimated for each treatment group are reported.
Time Frame: From the start of treatment to the date of first documentation of irPD, or date of death, whichever occurred first up to 1 year 6 months
Population: MITT included all participants enrolled and randomized to treatment and had an efficacy evaluation.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Denileukin Diftitox on Days 1 to 4 | Denileukin Diftitox on Days 1, 8, and 15
Number analyzed (Participants) | 42 | 32
weeks | 12.1 [11.6 to 14.0] | 12.1 [11.6 to 13.0]

3. Secondary Outcome: Percentage of Participants With PFS at Month 6
Description: The PFS was defined as time from start of study treatment until irPD or death. If the participant did not progress, the participant was censored at the date of last tumor assessment, known alive, or until starting a next line of therapy, whichever occurred first. PFS was assessed by irRC. irPD was defined as at least 25% increase in tumor burden relative to nadir (at any single time point) in 2 consecutive observations at least 4 weeks apart. Percentage of participants with PFS at month 6 are reported and was estimated using the Kaplan-Meier method.
Time Frame: Month 6
Population: MITT included all participants enrolled and randomized to treatment and had an efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Denileukin Diftitox on Days 1 to 4 | Denileukin Diftitox on Days 1, 8, and 15
Number analyzed (Participants) | 42 | 32
percentage of participants | 28.5 [15.2 to 43.3] | 23.0 [9.7 to 39.6]

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from date of the first assessment demonstrating an irCR or irPR to date of the first assessment demonstrating progressive disease (PD), death, or withdrawal from study. In the absence of confirmation of death or PD, duration of response was censored at the last date of follow-up when the participant was known to be alive and have maintained a response. Duration of response was assessed by irRC. Per irRC criteria, irCR was defined as complete disappearance of all tumor lesions, whether measurable or not, and no new lesions. irPR was defined as decrease in tumor burden by 50% or greater (confirmed in 2 observations at least 4 weeks apart). The duration of response was estimated using the Kaplan-Meier method.
Time Frame: From date of the first demonstration of irCR or irPR until the date of first demonstration of PD, date of death, or withdrawal from study up to 1 year 6 months
Population: MITT included all participants enrolled and randomized to treatment and had an efficacy evaluation. Here "overall number of participants analyzed" signifies participants who had confirmed irCR or irPR.
Measure: Median (Full Range); unit: weeks
Arm/Group | Denileukin Diftitox on Days 1 to 4 | Denileukin Diftitox on Days 1, 8, and 15
Number analyzed (Participants) | 4 | 1
weeks | 32.9 [26.6 to 49.6] | 54.3 [54.3 to 54.3]

5. Secondary Outcome: Overall Survival (OS)
Description: The OS was defined as the time from the date of randomization until the date of death. OS was estimated by Kaplan-Meier method. The median time (weeks) and the corresponding 90% confidence interval were estimated for each treatment group were reported.
Time Frame: From the date of randomization until the date of death up to 1 year 6 months
Population: MITT included all participants enrolled and randomized to treatment and had an efficacy evaluation.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Denileukin Diftitox on Days 1 to 4 | Denileukin Diftitox on Days 1, 8, and 15
Number analyzed (Participants) | 42 | 32
weeks | 51.1 [37.1 to 113.6] | 54.3 [30.7 to 77.1]

6. Secondary Outcome: Percentage of Participants With OS at 1 Year
Description: The OS was defined as the time from the date of randomization until the date of death. OS at 1 year was estimated by Kaplan-Meier method. OS at 1 year was measured as the percentage of participants still alive at 1 year from the date of randomization.
Time Frame: From the date of randomization up to 1 year
Population: MITT included all participants enrolled and randomized to treatment and had an efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Denileukin Diftitox on Days 1 to 4 | Denileukin Diftitox on Days 1, 8, and 15
Number analyzed (Participants) | 42 | 32
percentage of participants | 42.8 [21.9 to 62.3] | 50.0 [29.0 to 67.7]

7. Secondary Outcome: Change From Baseline in CD4+CD127-/loCD25+CD152- Cells Expression Pattern at Weeks 12
Description: Treg (regulatory T cells) from peripheral blood and tumor tissues were assessed for best immune-related response. Assessment of Treg cells was done by immunohistochemical (IHC) analysis. Change from baseline in CD4+CD127-/loCD25+CD152- (surface marker expressed in Treg cells) expression pattern, by treatment and immune-related response are reported.
Time Frame: Baseline, Week 12
Population: MITT included all participants enrolled and randomized to treatment and had an efficacy evaluation. Here 'N' (overall number of participants analyzed) included all participants who were evaluable for this outcome measure and 'n' (number analyzed) included all participants who were evaluable at specified timepoints for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells per microliter
Arm/Group | Denileukin Diftitox on Days 1 to 4 | Denileukin Diftitox on Days 1, 8, and 15
Number analyzed (Participants) | 39 | 29
cells per microliter
  At Baseline | 135.9 (86.17) | 184.9 (114.90)
  Change at Week 12: number analyzed (Participants) | 29 | 26
  Change at Week 12 | 6.4 (69.63) | -46.1 (74.72)

8. Secondary Outcome: Change From Baseline in CD4+CD127-/loCD25hiCD152- Cells Expression Pattern at Weeks 12
Description: Treg (regulatory T cells) from peripheral blood and tumor tissues were assessed for best immune-related response. Assessment of Treg cells was done by IHC analysis. Change from baseline in CD4+CD127-/loCD25hiCD152- (surface marker expressed in Treg cells) expression pattern, by treatment and immune-related response are reported.
Time Frame: Baseline, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells per microliter
Arm/Group | Denileukin Diftitox on Days 1 to 4 | Denileukin Diftitox on Days 1, 8, and 15
Number analyzed (Participants) | 39 | 29
cells per microliter
  At Baseline | 34.8 (16.58) | 40.0 (21.01)
  Change at Week 12: number analyzed (Participants) | 29 | 26
  Change at Week 12 | -8.0 (19.22) | -13.3 (13.37)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to approximately 1 year 6 months
Arm/Group | Denileukin Diftitox on Days 1 to 4 | Denileukin Diftitox on Days 1, 8, and 15
All-Cause Mortality (participants affected / at risk) | 22/43 | 17/32
Serious Adverse Events (participants affected / at risk) | 15/43 | 8/32
Other Adverse Events (participants affected / at risk) | 43/43 | 9/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denileukin Diftitox on Days 1 to 4 (N=43) | Denileukin Diftitox on Days 1, 8, and 15 (N=32)
Atrial Tachycardia (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Generalised Oedema (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Endocarditis Bacterial (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain Oedema (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 2 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denileukin Diftitox on Days 1 to 4 (N=43) | Denileukin Diftitox on Days 1, 8, and 15 (N=32)
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Vitreous floaters (Eye disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Nausea (Gastrointestinal disorders) | 24 | 4
Vomiting (Gastrointestinal disorders) | 9 | 1
Asthenia (General disorders) | 3 | 0
Chills (General disorders) | 20 | 3
Fatigue (General disorders) | 25 | 1
Generalised oedema (General disorders) | 3 | 0
Influenza like illness (General disorders) | 3 | 1
Pain (General disorders) | 4 | 0
Pyrexia (General disorders) | 6 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 2
Alanine aminotransferase increased (Investigations) | 12 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (Nervous system disorders) | 4 | 2
Dysgeusia (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 7 | 1
Restless legs syndrome (Nervous system disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 8 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 0
Hypotension (Vascular disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No